CLINICAL TRIAL: NCT01926899
Title: A Multicenter Phase I Study Evaluating the Addition of Bortezomib to an Established Acute Graft Versus Host Disease (aGVHD) Prophylaxis Regimen in Pediatric Allogeneic Hematopoietic Stem Cell Transplant (Allo HSCT) Patients
Brief Title: A Multicenter Phase I Study Evaluating the Addition of Bortezomib to an Established Acute Graft Versus Host Disease Prophylaxis Regimen in Pediatric Allogeneic Hematopoietic Stem Cell Transplant Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, David Delgado, Clinical Director of Pediatric Stem Cell Transplant, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1209009655
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Hematopoetic Stem Cell Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib administration (Experimental): 0.7 milligrams per meter squared given on Day 0 and Day +3
  Interventions: Drug: Bortezomib administration

INTERVENTIONS:
Drug: Bortezomib administration

SUMMARY:
The objective of this study is to determine the maximum tolerated dose (MTD) of bortezomib in combination with calcineurin inhibitor and methotrexate as acute graft versus host disease (aGVHD) prophylaxis in pediatric patients undergoing allogeniec hematopoietic stem cell transplant (alloHSCT)

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

  * Female subject of childbearing potential agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agree to completely abstain from heterosexual intercourse.
  * Male subjects, even if surgically sterilized (i.e., status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.
  * Subjects must be greater than or equal to 1 years old and less 22 years old.
  * Subjects must have any malignant or non-malignant condition that requires treatment with alloHSCT
  * Karnofsky or Lansky performance score greater than 60%
  * Subjects must have a 9 of 10 (HLA A, B, C, DR, and DQ) or 10 of 10 HLA matched-related or MUD for bone marrow or peripheral blood alloHSCT
  * Subjects must meet other institutional criteria for alloHSCT

Exclusion Criteria:

* • Patient has greater than 1.5 times upper limit normal (ULN) Total Bilirubin

  * Patient has greater than or equal to Grade 2 peripheral neuropathy
  * Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
  * Patient has hypersensitivity to bortezomib, boron, or mannitol.
  * Female subject is pregnant or lactating. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for postmenopausal or surgically sterilized women.
  * Female patients who are lactating or have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on Day 1 before first dose of study drug, if applicable.
  * Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
  * Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
  * Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
  * Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
  * Current active infection per physician determination
  * HIV positive
  * Previous myeloablative autoHSCT or alloHSCT in previous 12 months
  * ALT and AST greater than 5 times ULN for age
  * Creatinine clearance or glomerular filtration rate (GFR) less than 60 ml/min/1.73
  * Shortening fraction less than 26% or ejection fraction less than 45%
  * Diffusing capacity of carbon monoxide (DLCO), volume exhaled at end of first second of forced expiration (FEV1), diffusion capacity less than 50% of predicted (corrected for hemoglobin); if unable to perform lung function tests, oxygen saturation less than 94% on room air

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bortezomib | 100 days post transplant

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Texas Transplant Institute, San Antonio, Texas